CLINICAL TRIAL: NCT01653262
Title: An Open-label, Multicenter, Single-arm Study to Evaluate the Reduction in Nonpsychotic Behavioral Side Effects in Subjects With Epilepsy Switching From Levetiracetam to Brivaracetam Due to Nonpsychotic Behavioral Side Effects Phase 3b
Brief Title: Effect of Brivaracetam (BRV) on Nonpsychotic Behavioral Side Effects in Subjects Treated Previously With Levetiracetam (LEV)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma SA (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01395; 2011-005177-23 (EudraCT Number)
Expanded Access: NCT03532516 (Available)
Record Dates: First submitted 2012-07-26; First posted 2012-07-30 (Estimated); Results first posted 2016-08-15 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2016-07

CONDITIONS: Epilepsy
Keywords: Brivaracetam; Levetiracetam; Epilepsy; Nonpsychotic behavior
MeSH Terms: conditions — Epilepsy | interventions — brivaracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brivaracetam (Experimental): The subjects will be treated with Brivaracetam (BRV) tablets 200 mg/day during 12 weeks: four 25 mg tablets, twice daily.
  Based on the Investigator's judgement, at any time, the dose can be decreased to BRV 150 mg/day, 100 mg/day, or 50 mg/day. Flexible dosing, can be up- and down-titrated as needed.
  At the end of the Treatment Period, the subject will either enter the N01372 long-term follow-up study or down-titrate during 4 weeks.
  Interventions: Drug: Brivaracetam

INTERVENTIONS:
Drug: Brivaracetam

SUMMARY:
Trial N01395 is to evaluate the reduction of nonpsychotic behavioral side effects in subjects with Epilepsy who switched to BRV 200 mg/day after discontinuing LEV due to such side effects; as well as the efficacy, safety and tolerability of BRV. No statistical hypothesis testing will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Subject with well-characterized Epilepsy according to the 1989 International League Against Epilepsy (ILAE) classification
* Subject with Epilepsy who the investigator expects will benefit from Levetiracetam (LEV) but for whom the investigator has decided to discontinue due to nonpsychotic behavioral side effects following the introduction of LEV
* Subject is currently receiving LEV at the recommended therapeutic dose (dose ranging from 1 g/day to 3 g/day)
* Subject currently treated with minimum 2 and maximum 3 Anti-Epileptic Drugs (AEDs) including LEV. Vagal Nerve Stimulation (VNS) is allowed and will be counted as a concomitant AED
* Female subjects without childbearing potential (postmenopausal for at least 2 years, bilateral oophorectomy or tubal ligation, complete hysterectomy) are eligible. Female subjects with childbearing potential are eligible if they use a medically accepted contraceptive method

Exclusion Criteria:

* Subject has a lifetime history of suicide attempt (including an actual, interrupted or aborted attempt), or has had suicidal ideation in the past 6 months as indicated by a positive response ("Yes") to either Question 4 or Question 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS) at Visit 1
* Subject whose seizures could not be reliably counted on a regular basis due to their fast and repetitive occurrence (clusters or flurries)
* Subject has history or presence of status epilepticus during the year preceding Visit 1 or during Baseline
* Subject has history or presence of known psychogenic nonepileptic seizures
* Subject has any clinical conditions (eg, bone marrow depression, chronic hepatic disease, and/or severe renal impairment) which impair reliable participation in the study or necessitate the use of medication not allowed by protocol
* Subject is pregnant or lactating

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-07; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (12):
- United States (6):
  - 103, Little Rock, Arkansas
  - 108, Lexington, Kentucky
  - 109, New York, New York
  - 106, Akron, Ohio
  - 110, Dallas, Texas
  - 102, Salt Lake City, Utah
- France (2):
  - 203, Amiens
  - 201, Paris
- Germany (2):
  - 303, Bernau
  - 300, Kehl-Kork
- 502, Seville, Spain
- 603, Salford, United Kingdom

REFERENCES:
- [Derived] Yates SL, Fakhoury T, Liang W, Eckhardt K, Borghs S, D'Souza J. An open-label, prospective, exploratory study of patients with epilepsy switching from levetiracetam to brivaracetam. Epilepsy Behav. 2015 Nov;52(Pt A):165-8. doi: 10.1016/j.yebeh.2015.09.005. Epub 2015 Sep 29. PMID 26432008

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study started to enroll subjects in July 2012. In Oct 2013, the Sponsor evaluated the study in light of the recruitment rate. Given the unanticipated lack of recruitment during the prior 8 weeks, a decision was made to stop recruitment as of 16 Oct 2013.
Pre-assignment Details: Participant Flow refers to the Enrolled Set. In total, 32 subjects were screened and 29 subjects were enrolled instead of 30 subjects as per protocol amendment 2. This difference was considered as insignificant and not affecting the planned analysis.
Period: Overall Study
Arm/Group | Brivaracetam
Started | 29
Completed | 26
Not Completed | 3
Not completed — Lack of Efficacy | 1
Not completed — SAE, non-fatal | 1
Not completed — AE, non-serious non-fatal | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Enrolled Set.
Arm/Group | Brivaracetam
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.8 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Achieved a Clinically Meaningful Reduction of Nonpsychotic Behavioral Side Effects Based on the Investigator's Overall Assessment From Study Entry to the End of the Treatment Period
Description: Nonpsychotic behavioral side effects include (but are not limited to) such symptoms as aggression, agitation, anger, anxiety, apathy, depersonalization, depression, emotional lability, hostility, irritability, etc.
  The Investigator completed the assessment by answering the following:
  "Has there been a clinically meaningful reduction of nonpsychotic behavioral side effects since the start of BRV?"
  - Yes/No
Time Frame: From Study Entry (Visit1, Week -1) to the end of the Treatment Period (Visit 6, Week 12) or Early Discontinuation Visit
Population: The Full Analysis Set (FAS) consisted of all subjects who received at least 1 dose of Brivaracetam and had at least 1 post-Baseline evaluation of behavioral side effects.
Measure: Number; unit: percentage of subjects
Arm/Group | Brivaracetam
Number analyzed (Participants) | 29
percentage of subjects | 93.1

2. Secondary Outcome: Shift in the Maximum Intensity From Baseline to the End of the Treatment Period for Side Effects Primarily Associated With Discontinuation of Levetiracetam (LEV) as Determined by the Investigator
Description: Nonpsychotic behavioral side effects include (but are not limited to) such symptoms as aggression, agitation, anger, anxiety, apathy, depersonalization, depression, emotional lability, hostility, irritability, etc.
Time Frame: From Baseline (maximum of 12 weeks prior to Study Entry at Week -1) to the end of the Treatment Period (Visit 6, Week 12) or Early Discontinuation Visit
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Brivaracetam
Number analyzed (Participants) | 29
subjects
  Improvement | 8
  Unchanged | 2
  Worsening | 0
  Resolved | 19

3. Secondary Outcome: Change From Study Entry in Nonpsychotic Behavioral Side Effects to the End of the Treatment Period/Early Discontinuation Visit, Measured by Means of the Investigator Global Evaluation of Nonpsychotic Behavioral Side Effects (I-GEBSE) Scale
Description: There are seven levels for the I-GEBSE:
  * Marked improvement
  * Moderate improvement
  * Slight improvement
  * No change
  * Slight worsening
  * Moderate worsening
  * Marked worsening
Time Frame: From Study Entry (Visit1, Week -1) to the end of the Treatment Period (Visit 6, Week 12) or Early Discontinuation Visit
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Brivaracetam
Number analyzed (Participants) | 29
subjects
  Marked improvement | 10
  Moderate improvement | 10
  Slight improvement | 4
  No change | 2
  Slight worsening | 1
  Moderate worsening | 0
  Marked worsening | 1
  Missing | 1

4. Secondary Outcome: Number of Subjects Who Have a Complete Abatement of Nonpsychotic Behavioral Side Effects for the Last Assessment During the Treatment Period, Based on the Investigator's Overall Assessment
Description: as for outcome 2
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Brivaracetam
Number analyzed (Participants) | 29
subjects | 18

5. Secondary Outcome: Number of Subjects Who Are Free From Nonpsychotic Behavioral Side Effects Over the Entire Treatment Period
Description: Nonpsychotic behavioral side effects (NBSE) include (but are not limited to) such symptoms as aggression, agitation, anger, anxiety, apathy, depersonalization, depression, emotional lability, hostility, irritability, etc.
Time Frame: From Visit 2 (Week 0) to Visit 6 (Week 12)
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Brivaracetam
Number analyzed (Participants) | 29
subjects | 3

6. Secondary Outcome: Incidence of Treatment Emergent Adverse Events During the Study Period
Description: An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. A treatment emergent AE is any event that emerges during treatment having been absent pre-treatment, or worsens relative to the pre-treatment state.
Time Frame: From Study Entry (Visit1, Week -1) to the end of the Treatment Period (Visit 6, Week 12) or Early Discontinuation Visit
Population: The Safety Set (SS) consisted of all subjects who received at least 1 dose of Brivaracetam.
Measure: Number; unit: events
Arm/Group | Brivaracetam
Number analyzed (Participants) | 29
events | 67

7. Secondary Outcome: Withdrawal Due to an Adverse Event (AE) During the Study Period
Description: An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment.
Time Frame: From Study Entry (Visit1, Week -1) to the end of the Treatment Period (Visit 6, Week 12) or Early Discontinuation Visit
Population: The Safety Set (SS) consisted of all subjects who received at least 1 dose of Brivaracetam.
Measure: Number; unit: subjects
Arm/Group | Brivaracetam
Number analyzed (Participants) | 29
subjects | 2

8. Secondary Outcome: Occurrence of Serious Adverse Events During the Study Period
Description: A serious adverse event is any untoward medical occurrences in a subject administered study treatment, whether or not the event is related to treatment, with at least one of the follow outcomes: death, life-threatening, initial inpatient hospitalization or prolongation of hospitalization, significant or persistent disability/incapacity, congenital anomaly/birth defect, or an important medical event that may jeopardize the subject and require a medical/surgical intervention.
Time Frame: From Study Entry (Visit1, Week -1) to the end of the Treatment Period (Visit 6, Week 12) or Early Discontinuation Visit
Population: The Safety Set (SS) consisted of all subjects who received at least 1 dose of Brivaracetam.
Measure: Number; unit: events
Arm/Group | Brivaracetam
Number analyzed (Participants) | 29
events | 1

9. Secondary Outcome: Partial Onset Seizure (POS) Frequency Over the Treatment Period for Subjects With Focal Epilepsy
Description: The POS frequency is standardized to a 28-day duration and changes in POS frequency are measured relative to the reported seizure counts for the 4 weeks prior to Visit 2 (Week 0).
  Partial seizures can be classified into one of the following three groups:
  * Simple partial seizures (IA)
  * Complex partial seizures (IB)
  * Partial seizures evolving to secondarily generalized seizures (IC)
Time Frame: From 4 weeks prior to Visit 2 (Week 0) to the end of the Treatment Period (Visit 6, Week 12) or Early Discontinuation Visit
Population: The Efficacy Analysis Set (EAS) consisted of all subjects who received at least 1 dose of Brivaracetam and had at least 1 post-Baseline day of seizure daily record card (subject diary card).
Measure: Median (Inter-Quartile Range); unit: partial onset seizures
Arm/Group | Brivaracetam
Number analyzed (Participants) | 15
partial onset seizures | 6.0 [2.2 to 17.7]

10. Secondary Outcome: Generalized Seizure Days Over the Treatment Period for Subjects With Idiopathic Generalized Epilepsy
Description: Generalized seizure days are standardized to a 28-day duration and changes in generalized seizure days are measured relative to the reported seizure counts for the 4 weeks prior to Visit 2 (Week 0).
  Generalized seizures (Type II) include the following seizure types:
  * Absence (IIA1)
  * Atypical absence (IIA2)
  * Myoclonic (IIB)
  * Clonic (IIC)
  * Tonic (IID)
  * Tonic-clonic (IIE)
  * Atonic (IIF)
  A specific effect of BRV on the occurrence of generalized seizures was not assessed.
Time Frame: as for outcome 9
Population: This variable was not analyzed and no results are available.
Arm/Group | Brivaracetam
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from Screening Period (Week -1) over the 12-weeks Treatment Period until the Safety Visit (Week 15-18 + max 7 days).
Description: Adverse Events refer to the Safety Set (SS) consisting of all subjects who received at least 1 dose of Brivaracetam.
Arm/Group | Brivaracetam
Serious Adverse Events (participants affected / at risk) | 1/29
Other Adverse Events (participants affected / at risk) | 13/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brivaracetam (N=29)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brivaracetam (N=29)
Fatigue (General disorders) | 3 (3)
Nasopharyngitis (Infections and infestations) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Headache (Nervous system disorders) | 5 (7)
Dizziness (Nervous system disorders) | 2 (2)
Tremor (Nervous system disorders) | 2 (2)
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days